### **Research Study Informed Consent Document**

Study Title for Study Participants: Implementation of Smoking Cessation Services (OaSiS)

Official Study Title for Internet Search on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>: Implementation of Smoking Cessation Services within NCI NCORP Community Sites with Organized Lung Cancer Screening Program (NCT03291587)

Informed Consent Form to Participate in Research for <u>Key Informant</u>

Site Principal Investigator

#### Introduction

You are being invited to take part in a research study. This study has public funding from the National Cancer Institute (NCI), part of the National Institutes of Health (NIH) in the United States Department of Health and Human Services. Your participation is voluntary. You do not have to participate in this study. There is no penalty for choosing not to participate.

Why is this study being done? We are evaluating a training program to help lung cancer screening clinics improve their ability to support patients to quit smoking. We are conducting this study in 26 clinics, half of the clinics receive the training and the other half do not. Our goal is to determine if our training program helps the clinic improve their services.

## Why are these interviews being done?

We are conducting these interviews because we want to learn what health professionals think about the implementation of evidence-based tobacco cessation strategies in community-based lung cancer screening facilities. We are inviting key informants at participating screening programs to participate at the beginning and after implementation of the intervention. We plan to conduct interviews with three personnel at each site. Each participant will be interviewed once at the beginning of the study and once near completion of the study. We expect to enroll 78 participants. Participating in an interview will not give you any direct benefits, but we hope the information we learn will help health professionals in the future to determine the most feasible and appropriate cessation strategies for lung cancer imaging facilities.

#### What is involved?

A study interviewer will meet with you by telephone for approximately 30 minutes at a time that is convenient for you. The interviewer will ask you questions about the clinic's current cessation support services, the feasibility and appropriateness of offering various cessation services, and the potential opportunities and challenges for implementing these services in your clinic. You will receive a \$25 gift card as a thank-you for your time.

# How long will I be in this study?

The duration of this study is planned for 4.5 years. You will be interviewed twice during the study.

#### What possible risks can I expect from taking part in this study?

Your participation in this research will only concern routine, every-day professional behaviors related to tobacco cessation services in relation to an organized cancer screening program, in the course of daily work. No personal information will be requested. Efforts, such as coding research records, keeping research records secure and allowing only authorized people to have access to research records, will be made to keep your information safe.

We will audio-record the interviews for later analysis by the research team, and we will remove your name from the transcribed version. We want to protect your privacy, so we will not use your name or any identifying information in any report we might publish. Your participation is voluntary, and you may choose to stop participating at any time without penalty. We will destroy the audio recordings once this study is finished. There may be some risks that the study team does not yet know about.

### What possible benefits can I expect from taking part in this study?

Participating in an interview will not give you any direct benefits, but we hope the information we learn will help health professionals and patients in the future.

### Can I stop taking part in this study?

Yes, you can decide to stop at any time. If you decide to stop for any reason, we ask that you let the study staff person know as soon as possible.

### What are my rights in this study?

Taking part in this study is voluntary. If for some reason you decide not to participate, this will in no way affect your role/work as a member of the staff of the screening facility. For questions about your rights while in this study, call the (insert local IRB) at (insert telephone number).

## What are the costs of taking part in this study?

There are no costs to you for taking part in this study.

You will receive a \$25 gift card as a thank-you for your time.

## Where can I get more information?

You may visit the NCI Web site at <a href="http://cancer.gov/">http://cancer.gov/</a> for more information about studies or general information about cancer. You may also call the NCI Cancer Information Service to get the same information at: 1-800-4-CANCER (1-800-422-6237).

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## Who can answer my questions about this study?

You can talk to study staff about any questions or concerns you have about this study. If you later have questions, you may contact the study investigators *Site Contact Information Here*.

# My Signature Agreeing to Take Part in the Study

I have read this consent form or had it read to me. I have discussed it with the study doctor and my questions have been answered. I will be given a signed copy of this form. I agree to take part in the study.

| Participant's signature | | |
|---|---|---|
| Date of signature | Time of signature: | AM/PM |
| Signature of person(s) conducting the informed consent discussion | | |
| Date of signature | Time of signature: | AM/PM |